CLINICAL TRIAL: NCT02450539
Title: A Randomized Phase 2 Study of Abemaciclib (LY2835219) Versus Docetaxel in Patients With Stage IV Squamous Non-Small Cell Lung Cancer Previously Treated With Platinum-Based Chemotherapy
Brief Title: A Study of Abemaciclib (LY2835219) in Participants With Stage IV Squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15806; I3Y-MC-JPBX (Other: Eli Lilly and Company); 2014-004832-20 (EudraCT Number)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07-15

CONDITIONS: Non-Small Cell Lung Cancer Stage IV
Keywords: patient reported outcomes (PRO); patient focused outcomes (PFO); biomarkers; CDK 4 and 6
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abemaciclib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abemaciclib (Experimental): 200 milligram (mg) abemaciclib given orally every 12 hours (Q12H) on days 1 to 21 of each 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib
- Docetaxel (Active Comparator): 75 milligram per meter squared (mg/m²) docetaxel given intravenously (IV) on day 1 of each 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib
Drug: Docetaxel — Administered IV
  Arms: Docetaxel

SUMMARY:
The main purpose of this study is to evaluate the effectiveness of the study drug known as abemaciclib versus docetaxel in participants with stage IV squamous non-small cell lung cancer (NSCLC) previously treated with platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of stage IV NSCLC.
* Have progressed during or after platinum-based chemotherapy for advanced disease.
* Have not received prior treatment with docetaxel.
* Have availability of adequate formalin-fixed paraffin-embedded (FFPE) tumor derived material.
* Have adequate organ function including hematology, renal, and liver.
* Have good performance score (0-1).
* Have measurable disease per RECIST 1.1.
* Agree to use a reliable medically approved method of birth control.

Exclusion Criteria:

* Have received prior treatment with any cyclin dependent kinase (CDK) 4 and 6 inhibitor or participated in a clinical trial with a CDK 4 and 6 inhibitor and the treatment administered is not known.
* Are currently receiving treatment in a clinical trial involving an investigational product or non-approved use of a drug or device.
* Have the presence of unstable central nervous system (CNS) metastasis.
* Have had major surgery (excluding biopsy) < 28 days of the initial dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-08-06 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (49):
- United States (5):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Washington University School of Medicine, St Louis, Missouri
  - Montefiore Medical Center, The Bronx, New York
  - Vista Oncology Inc. PS, Olympia, Washington
- Australia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Camperdown
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Randwick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Brisbane
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woolloongabba
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suresnes
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cologne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gera
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heidelberg
- Hungary (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Győr
- Italy (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olsztyn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
- Russia (2):
  - St-Petersburg scientifical practical center of specialized kinds of medical care (oncological), Saint Petersburg
  - Volgograd regional clinical oncology dispensary, Volzhsky
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cheongju-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulsan
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taichung
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- Ukraine (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kryvyi Rih
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnitsa

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Abemaciclib (LY2835219) in Participants With Stage IV Squamous Non-small Cell Lung Cancer — https://trials.lillytrialguide.com/en-US/trial/3fFmhLPCZ2EGMW8w6gCq0Y?conditionId=WWF5j0kxgqI0QYaYMo04G

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study completers are participants who died due to any cause, were on follow-up at study completion or completed continued access period.
Groups:
- Abemaciclib: 200 milligram(mg) abemaciclib given orally every 12 hours (Q12H) on days 1 to 21 of each 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Abemaciclib | Docetaxel
Started | 106 | 53
Received at Least One Dose of Study Drug | 106 | 52
Completed | 90 | 46
Not Completed | 16 | 7
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abemaciclib | Docetaxel | Total
Number analyzed (Participants) | 106 | 53 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (7.8) | 64.5 (7.1) | 63.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 90 | 44 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 84 | 48 | 132
  Unknown or Not Reported | 17 | 2 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 3 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 96 | 50 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 18 | 4 | 22
  Hungary | 7 | 6 | 13
  United States | 4 | 2 | 6
  Ukraine | 13 | 13 | 26
  Russia | 11 | 2 | 13
  Spain | 8 | 6 | 14
  South Korea | 8 | 1 | 9
  Taiwan | 2 | 2 | 4
  Poland | 14 | 10 | 24
  Italy | 7 | 1 | 8
  Australia | 4 | 0 | 4
  France | 1 | 2 | 3
  Germany | 9 | 4 | 13
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were stratified at randomization according to the following: Eastern Cooperative Oncology Group (ECOG) PS (0 vs. 1); number of prior therapies (received only platinum-based therapy vs. platinum-based therapy plus immune checkpoint inhibitor) and time since initiation of first line therapy (<=9 months vs >9 months). The ECOG Performance Status:0 - Fully active, able to carry on all pre-disease performance without restriction,1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Participants
    0 | 22 | 7 | 29
    1 | 84 | 46 | 130

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from the date of randomization to the date of investigator-determined disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) or death from any cause. Progressive disease (PD) was defined as at least a 20% increase in the sum of the longest diameters (LD) of target lesions, with reference the smallest sum on study and an absolute increase of at least 5mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant was not known to have died or have objective progression, PFS time will be censored at the day of their last radiographic tumor assessment (if available) or date of randomization if no post baseline radiographic assessment is available.
Time Frame: Baseline to Objective Progression or Death from Any Cause ( Up To 6 Months)
Population: All participants according to the treatment group to which they were randomized. Participants censored: Abemaciclib=19 and Docetaxel= 15.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib | Docetaxel
Number analyzed (Participants) | 106 | 53
months | 2.53 [1.68 to 2.89] | 4.21 [2.79 to 5.65]
Statistical Analysis 1: Comparison: Abemaciclib vs Docetaxel; Stratified by baseline ECOG performance status (0 vs 1), number of Prior Therapies (received only platinum-based therapy vs Received platinum-based Therapy plus Immune Checkpoint Inhibitor), and time since initiation of first line therapy (<=9 months vs >9 months); Test type: Superiority; p = 0.0068, Stratified log-rank test; Hazard Ratio (HR) = 1.765, 95% CI 2-sided [1.165 to 2.672] — Stratified Cox proportional hazard model

2. Secondary Outcome: Pharmacokinetics (PK): Clearance of Abemaciclib
Description: Pharmacokinetics (PK): Clearance of Abemaciclib
Time Frame: Cycle (C) 1 Day (D) 1: Pre-dose; C1D8: 4 and 7 hr Post-dose; C2D1: Pre-dose and 3 hr Post-dose; C3 and C4 D1:Pre-dose
Population: All participants who received abemaciclib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hour (L/h)
Groups:
- Abemaciclib: 200 milligram(mg) abemaciclib given orally every 12 hours (Q12H) on days 1 to 21 of each 21 day cycle.
Arm/Group | Abemaciclib
Number analyzed (Participants) | 102
Liters/hour (L/h) | 21.3 (36)

3. Secondary Outcome: PK: Volume of Distribution of Abemaciclib
Description: PK: Volume of Distribution of Abemaciclib
Time Frame: Cycle (C) 1 Day (D) 1: Pre-dose; C1D8: 4 and 7 hr Post-dose; C2D1: Pre-dose and 3 hr Post-dose; C3 and C4 D1:Pre-dose
Population: All participants who received Abemaciclib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Abemaciclib
Number analyzed (Participants) | 102
Liters (L) | 769 (51)

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death due to any cause. For each participant who is not known to have died as the data inclusion cutoff date for overall survival analysis, OS time was censored on the last date the participant is known to be alive.
Time Frame: Baseline to Date of Death from Any Cause (Up To 28 Months)
Population: All participants according to the treatment group to which they were randomized. Participants censored: Abemaciclib=35 and Docetaxel= 17.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib | Docetaxel
Number analyzed (Participants) | 106 | 53
Months | 7 [5.00 to 8.78] | 12.39 [7.13 to 15.98]
Statistical Analysis 1: Comparison: Abemaciclib vs Docetaxel; Stratified by baseline ECOG performance status (0 vs 1), number of Prior Therapies (received only platinum-based therapy vs Received platinum-based Therapy plus Immune Checkpoint Inhibitor), and time since initiation of first line therapy (<=9 months vs >9 months).]; Test type: Superiority; p = 0.1746, Stratified log-rank test; Hazard Ratio (HR) = 1.333, 95% CI 2-sided [0.879 to 2.022] — Stratified Cox proportional hazard model

5. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR])
Description: Overall response was defined as the percentage of randomized participants achieving a best overall response (BoR) of complete response (CR) or partial response (PR) using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) criteria. Participants with unevaluable or unknown response status are considered nonresponders. Complete response (CR) is defined as the disappearance of all target and non-target lesions and no appearance of new lesions. Partial response (PR) is defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions and no appearance of new lesions.
Time Frame: Baseline to Objective Progression (Up To 6 Months)
Population: All randomized participants.
Measure: Number; unit: percentage participants
Arm/Group | Abemaciclib | Docetaxel
Number analyzed (Participants) | 106 | 53
percentage participants | 2.8 | 20.8
Statistical Analysis 1: Comparison: Abemaciclib vs Docetaxel; Test type: Superiority; Rate Difference = -17.9, 95% CI 2-sided [-29.3 to -6.6] — Confidence intervals are based on the normal approximation to the binomial

6. Secondary Outcome: Percentage of Participants Who Exhibit Stable Disease (SD) or Confirmed Response (CR) or Partial Response (PR): Disease Control Rate (DCR)
Description: DCR is the percentage of randomized participants who achieved a complete response, partial response or stable disease using Response Evaluation Criteria In Solid Tumors (RECIST v1.1) criteria. Complete response (CR) is defined as the disappearance of all target and non-target lesions, and no appearance of new lesions. Partial response (PR) is defined as at least a 30% decrease in the sum of longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions and no appearance of new lesions. Stable disease was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Baseline through Measured Progressive Disease or Death Due to Any Cause (Up To 6 Months)
Population: All randomized participants.
Measure: Number; unit: percentage participants
Arm/Group | Abemaciclib | Docetaxel
Number analyzed (Participants) | 106 | 53
percentage participants | 50.9 | 64.2
Statistical Analysis 1: Comparison: Abemaciclib vs Docetaxel; Test type: Superiority; Rate Difference = -13.2, 95% CI 2-sided [-29.2 to 2.8] — Confidence intervals are based on the normal approximation to the binomial

7. Secondary Outcome: Time to Worsening of Eastern Cooperative Oncology Group (ECOG) Performance Status of >/=2
Description: Worsening of ECOG performance status is the duration from randomization to ECOG PFS of >/=2. Participants without an ECOG PFS >/=2 are censored at last adequate post baseline ECOG Performance Status or randomization date (whichever is last).
  The ECOG Performance Status:0 - Fully active, able to carry on all pre-disease performance without restriction,1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, 2 - Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours,3 - Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours, 4 - Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair, 5 - Dead
Time Frame: Randomization to ECOG PFS of >/=2 (Up To 11.5 Months)
Population: All randomized participants. Participants censored: Abemaciclib =93 and Docetaxel= 43.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib | Docetaxel
Number analyzed (Participants) | 106 | 53
months | NA [6.58 to NA] — Due to insufficient data to support the analysis and the results. | 10.52 [4.64 to NA] — Due to insufficient data to support the analysis and the results.
Statistical Analysis 1: Comparison: Abemaciclib vs Docetaxel; Stratification factors are baseline ECOG performance status (0 vs 1), Number of Prior Therapies (received only platinum-based therapy vs Received platinum-based Therapy plus Immune Checkpoint Inhibitor), and time since initiation of first line therapy (<=9 months vs >9 months); Test type: Superiority; p = 0.7039, Stratified Log Rank; Hazard Ratio (HR) = 1.184, 95% CI 2-sided [0.502 to 2.792] — Stratified Cox regression model

8. Secondary Outcome: Change From Baseline in MD Anderson Symptom Inventory-Lung Cancer (MDASI-LC) Scores
Description: MDASI-LC included 33 items:6 interference and 27 symptom(3 lung-cancer (LC),8 brain tumor (BT),and 3 study-specific(headache,diarrhea, and rash).Analyzed endpoints were 9 constructs:3 single-items (headache,diarrhea,and rash) and 6 composites(interference+core,LC,core+LC,BT, and core+LC worst 5 baseline).Data for all 9 constructs were collected by an 11-point numeric rating scale anchored at 0(not present or does not interfere) and 10(as bad as you can imagine or interfered completely).The measurement range was 10 (maximum score-minimum score). Between-group difference in regression-predicted change from baseline were estimated for each specified construct. MMRM models included independent variables treatment,visit, treatment*visit,and baseline score. Group-level negative change from baseline indicated group improvement.
Time Frame: Baseline through End of Study (Up To 6 Months)
Population: All randomized participants for cycles which at least 25% of participants in each arm have a score.MDASI-LC population included all randomized participants who completed at least 1 baseline assessment followed by at least 1 MDASI-LC assessment after Cycle 1 (for example, a completed MDASI-LC questionnaire at Cycle 2 Day 1 or later)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Abemaciclib | Docetaxel
Number analyzed (Participants) | 87 | 43
units on a scale
  Headache | 0.19 (0.14) | 0.01 (0.18)
  Diarrhea | 1.01 (0.18) | 0.15 (0.23)
  Mean core symptom severity | 0.53 (0.14) | 0.00 (0.18)
  Mean interference | 0.50 (0.20) | 0.18 (0.27)
  Mean lung cancer symptom severity | 0.20 (0.12) | -0.19 (0.15)
  Mean core plus lung cancer symptom severity | 0.47 (0.13) | -0.04 (0.17)
  Mean brain tumor symptom severity | 0.19 (0.11) | 0.13 (0.15)
  Mean core plus lung worst 5 symptoms severity | -0.25 (0.17) | -0.94 (0.22)
  Rash | 0.28 (0.14) | 0.18 (0.17)
Statistical Analysis 1: Comparison: Abemaciclib vs Docetaxel; Headache; Test type: Superiority; Mean Difference (Final Values) = 0.18, Standard Error of Mean 0.23
Statistical Analysis 2: Comparison: Abemaciclib vs Docetaxel; Diarrhea; Test type: Superiority; Mean Difference (Final Values) = 0.86, Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Abemaciclib vs Docetaxel; Mean core symptom severity; Test type: Superiority; Mean Difference (Final Values) = 0.53, Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Abemaciclib vs Docetaxel; Mean interference; Test type: Superiority; Mean Difference (Final Values) = 0.32, Standard Error of Mean 0.34
Statistical Analysis 5: Comparison: Abemaciclib vs Docetaxel; Mean lung cancer symptom severity; Test type: Superiority; Mean Difference (Final Values) = 0.39, Standard Error of Mean 0.19
Statistical Analysis 6: Comparison: Abemaciclib vs Docetaxel; Mean core plus lung cancer symptom severity; Test type: Superiority; Mean Difference (Final Values) = 0.52, Standard Error of Mean 0.21
Statistical Analysis 7: Comparison: Abemaciclib vs Docetaxel; Mean brain tumor symptom severity; Test type: Superiority; Mean Difference (Final Values) = 0.06, Standard Error of Mean 0.19
Statistical Analysis 8: Comparison: Abemaciclib vs Docetaxel; Mean core plus lung worst 5 symptoms severity; Test type: Superiority; Mean Difference (Final Values) = 0.69, Standard Error of Mean 0.28
Statistical Analysis 9: Comparison: Abemaciclib vs Docetaxel; Rash; Test type: Superiority; Mean Difference (Final Values) = 0.09, Standard Error of Mean 0.22

9. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional 5-Level (EQ-5D-5L) Questionnaire EQ VAS Overall Self-rated Health Score
Description: The EQ-5D-5L is a standardized instrument for use as a measure of self-reported health status. Overall self-rated health was measured with a vertical 20 cm visual analog scale (VAS) anchored at 0 (worst health) and ranged through 100 (best health). Between-group differences in regression-predicted change from baseline score were estimated for VAS scores. MMRM models included independent variables treatment, visit, treatment*visit, and baseline score. Group-level negative change from baseline indicated group improvement.
Time Frame: Baseline to Measured Progressive Disease (Up To 6 Months)
Population: All randomized participants for cycles which at least 25% of participants in each arm have a score.The EQ-5D-5L population included all randomized participants who completed at least 1 baseline assessment followed by at least 1 EQ-5D-5L assessment after Cycle 1 (for example, a completed EQ-5D-5L questionnaire at Cycle 2 Day 1 or later).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Abemaciclib | Docetaxel
Number analyzed (Participants) | 88 | 42
units on a scale | -5.49 (1.28) | -2.36 (1.63)
Statistical Analysis 1: Comparison: Abemaciclib vs Docetaxel; EQ VAS Overall Self-rated Health Score; Test type: Superiority; Mean Difference (Final Values) = -3.13, Standard Error of Mean 2.07

10. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional 5-Level (EQ-5D-5L) Questionnaire Index Value
Description: There are 5 response levels on a good-to-bad continuum of 1-5 corresponding to none, slight, moderate, severe, and extreme/unable to.The EuroQol-developed crosswalk method was used to convert the EQ-5D-5L,using UK weights,health dimensions(mobility,self-care,usual activities,pain/discomfort, and anxiety/depression) into a single index value;the dimensions are not separately scored.The index is marked missing when ≥1 dimensions are missing.The index scores for the response patterns were anchored on full health to dead with negative values assigned to response patterns/health states considered worse than death.The best pattern is assigned the index value of 1.0; the worst pattern is assigned an index value of -0.594. Between-group differences in regression-predicted change from baseline score were estimated for the index .MMRM models included independent variables treatment, visit, treatment*visit, and baseline score.Group-level negative change from baseline indicated group improvement.
Time Frame: Baseline to Measured Progressive Disease (Up To 6 Months)
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Abemaciclib | Docetaxel
Number analyzed (Participants) | 88 | 42
units on a scale | -0.05 (0.02) | -0.01 (0.02)
Statistical Analysis 1: Comparison: Abemaciclib vs Docetaxel; EQ-5D-5L Index Value; Test type: Superiority; Median Difference (Final Values) = -0.04, Standard Error of Mean 0.03

ADVERSE EVENTS:
Time Frame: Baseline Up To 5 Years
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Abemaciclib | Docetaxel
All-Cause Mortality (participants affected / at risk) | 71/106 | 35/52
Serious Adverse Events (participants affected / at risk) | 29/106 | 17/52
Other Adverse Events (participants affected / at risk) | 94/106 | 43/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=106) | Docetaxel (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 6 (6) | 4 (4)
Myelitis (Infections and infestations) | 0 (0) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=106) | Docetaxel (N=52)
Anaemia (Blood and lymphatic system disorders) | 41 (47) | 12 (18)
Leukopenia (Blood and lymphatic system disorders) | 10 (10) | 14 (48)
Neutropenia (Blood and lymphatic system disorders) | 18 (20) | 26 (76)
Thrombocytopenia (Blood and lymphatic system disorders) | 27 (35) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 8 (10) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 41 (67) | 5 (5)
Nausea (Gastrointestinal disorders) | 33 (35) | 7 (10)
Vomiting (Gastrointestinal disorders) | 9 (11) | 3 (3)
Fatigue (General disorders) | 30 (34) | 7 (10)
Non-cardiac chest pain (General disorders) | 8 (9) | 2 (2)
Pain (General disorders) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 5 (5) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 3 (3)
Blood creatinine increased (Investigations) | 13 (17) | 1 (6)
Weight decreased (Investigations) | 12 (13) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 17 (19) | 7 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (10) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (9) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 10 (12) | 7 (8)
Dizziness (Nervous system disorders) | 8 (10) | 3 (3)
Headache (Nervous system disorders) | 7 (7) | 2 (2)
Neuropathy (Nervous system disorders) | 3 (3) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 6 (6)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (8)
Hypotension (Vascular disorders) | 8 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT02450539/Prot_002.pdf
  • Statistical Analysis Plan (2015-06-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT02450539/SAP_001.pdf